CLINICAL TRIAL: NCT00820040
Title: To Examine the Feasibility of Using Permacol® Surgical Implant in the Repair of Abdominal Wall Defects After Removal of Chronic Infect Prosthetic Mesh
Brief Title: Feasibility of Permacol Use in Infected Fields
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment due to strict eligibility criteria
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hern06R2
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Hernia
Keywords: Hernia; Contaminated Field; Mesh Removal; infected mesh removal
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Permacol (Experimental)
  Interventions: Device: acellular porcine dermal collagen mesh

INTERVENTIONS:
Device: acellular porcine dermal collagen mesh — porcine mesh for hernia repair/ abdominal wall reconstruction
  Other Names: Permacol

SUMMARY:
This pilot study is to examine the feasibility of using Permacol Surgical Implant in the repair of abdominal wall defects after removal of infected prosthetic mesh

ELIGIBILITY:
Inclusion Criteria:

* Have given written Informed Consent
* Be 18-85 years of age (inclusive)
* Have prosthetic mesh that is in proximity to an infected wound that has failed conservative management for at least 3 months, with mesh exposure and a draining wound, or that is in proximity to an abscess that requires operative intervention.
* Have a wound characterized by purulent discharge, positive gram stain or positive culture to document infection
* Be a candidate for surgical removal of infected mesh placed for repair of ventral/incisional hernias and concomitant abdominal wall reconstruction
* Have an ASA Score ≤3
* Have a body mass index (BMI) between 16.5 and 40 inclusive
* Be a candidate for anticipated primary approximation of skin/wound
* Have a life expectancy of at least 18 months
* Be willing to allow biopsy of implant if secondary wound opening is performed or spontaneous implant exposure occurs

Exclusion Criteria:

* Have loss of abdominal domain such that the operation would be impractical or would adversely effect respiratory or cardiovascular function to an unacceptable degree
* Have an enterocutaneous fistula in proximity to wound/mesh
* Be a candidate for emergency surgery that would make giving valid Informed Consent impractical
* Be currently taking part in another clinical study that conflicts with the current study
* Have known allergy to porcine collagen products
* Have active generalized peritonitis or intraperitoneal sepsis
* Have active necrotizing fasciitis
* Have active abdominal compartment syndrome
* Have active untreated metabolic or systemic illness
* Report unintentional weight loss >10% of body weight in the previous 90 days
* Have known collagen metabolism disorder.(e.g., Ehlers-Danlos syndrome)
* Have known altered immune response (e.g., HIV or other immunodeficiency disorder))
* Have chronic renal failure
* Have known active malignancy present
* Have history of systemic chemotherapy within previous 1 year
* Have lifetime history of radiation to the abdomen, pelvis or thorax
* Have inguinal or groin hernia as primary diagnosis
* Be currently pregnant or planning to become pregnant during study period
* Be unable to give valid informed consent or comply with required follow- up schedule
* Suffer from mental capacity sufficiently severe to make informed consent unobtainable

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Roth, MD, Principal Investigator — University of Kentucky
Locations (3):
- United States (3):
  - University of Kentucky, Lexington, Kentucky
  - Albany Medical College, Albany, New York
  - Greenville Hospital System, Greenville, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects diagnosed with infected prosthetic mesh who were scheduled to undergo planned removal of the mesh were assessed for potential study eligibility.
  Subjects needed to fulfill all inclusion criteria and no exclusion criteria to be enrolled into the study.
Pre-assignment Details: One subject was considered a screen failure due to undergoing chemotherapy for an active malignancy within a year prior to the screening visit.
Groups:
- Permacol: acellular porcine dermal collagen mesh: porcine mesh for hernia repair/ abdominal wall reconstruction after removal of infected prosthetic mesh
Period: Overall Study
Arm/Group | Permacol
Started | 10
Safety Evaluable Population | 8
Full Analysis Set | 8
Completed | 7
Not Completed | 3
Not completed — Death | 1
Not completed — Sponsor terminated study | 1
Not completed — Screen failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Permacol
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Weight [Mean (Standard Deviation); unit: lb] | 253.1 (55.92)
Height [Mean (Standard Deviation); unit: inches] | 70.0 (5.58)
BMI [Mean (Standard Deviation); unit: kg/m²] | 36.91 (7.812)
Employment Status [Number; unit: participants]
  Disability/Sick Leave | 4
  Full Time | 2
  Missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hernia Recurrence or Surgical Site Infection Requiring Wound Opening
Description: The primary objective of this study was hernia recurrence or surgical site infection as assessed by a CT scan 12 months following surgery.Hernia recurrence was defined as any abnormal abdominal protrusion, as assessed by 12 month CT. Surgical site infection requiring wound opening was defined as abscess formation or drainage that required surgical wound opening. Wound opening was defined as surgical entry into the wound.
Time Frame: 12 months
Population: Hernia recurrence and Surgical Site Infection Requiring Wound Opening for one subject could not be assessed due to death unrelated to the study device. The subject died 19 days post-operatively and therefore primary endpoints assessed at 12 month visit were reported as missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Permacol
Number analyzed (Participants) | 8
Participants
  No Hernia Recurrence or Surgical Site Infection Requiring Wound Opening | 7
  Missing | 1

2. Secondary Outcome: Subjects Having Permacol Implants Removed or Debrided After Implantation
Description: The secondary objective of this study was the incidence of Permacol™ surgical implant removal or debridement. Removal was defined as complete surgical excision of the implant. Debridement was defined as debridement or lavage of ≥10% of the visible implant surface area as subjectively assessed by the operating surgeon.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Permacol
Number analyzed (Participants) | 8
Participants
  None Reported | 8
  Reported | 0

3. Other Pre Specified Outcome: Physical and Other Examinations
Description: The SF-12v2 Health Survey® (12-question short form health survey) measure eight domains of health related quality of life, which is then aggregated to provide summary measure of the respondent's physical and mental health. Results of 12-month abdominal CT examination are summarized as a change from the baseline. The SF-12v2 Health Survey® is broken into physical health and mental health. Physical health is determined by: physical functioning, role-playing, bodily pain and general health. Mental health is determined by: vitality, social functioning, role-emotional and mental health. The general population mean of the United States is 50. When analyzing the results, the mean values of the study subjects are taken and compared to the general United States population. Each 10 points represent one standard deviation. A measure of one standard deviation (10 points) below the population mean (50) indicates significant function impairment.
Time Frame: 12-month post-procedure change from baseline
Population: At baseline eight subjects completed the questionnaire and at 12 months there were seven subjects who completed the questionnaire due to the death of one patient.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Permacol
Number analyzed (Participants) | 7
score on a scale
  Physical Functioning | 12.37 (16.292)
  Role Physical | 10.28 (7.271)
  Bodily Pain | 7.73 (14.194)
  General Health | -0.57 (6.953)
  Social Functioning | 8.90 (10.270)
  Role Emotional | 11.14 (16.000)
  Vitality | 2.81 (14.715)
  Mental Health | 4.92 (9.027)
  Physical Component Score | 7.96 (10.167)
  Mental Component Score | 5.42 (8.769)

4. Other Pre Specified Outcome: Physical and Other Examinations
Description: as for outcome 3
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Permacol
Number analyzed (Participants) | 8
score on a scale
  Physical Functioning | 37.39 (10.304)
  Role Physical | 37.36 (7.417)
  Bodily Pain | 39.69 (12.754)
  General Health | 44.52 (13.225)
  Social Functioning | 41.34 (12.352)
  Role Emotional | 35.49 (14.437)
  Vitality | 47.84 (11.075)
  Mental Health | 46.28 (10.814)
  Physical Component Score | 39.18 (8.947)
  Mental Component Score | 44.61 (9.849)

5. Other Pre Specified Outcome: Physical and Other Examinations
Description: as for outcome 3
Time Frame: 12-month post-procedure
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Permacol
Number analyzed (Participants) | 7
score on a scale
  Physical Functioning | 49.19 (11.130)
  Role Physical | 47.19 (12.422)
  Bodily Pain | 47.42 (12.134)
  General Health | 45.48 (12.223)
  Social Functioning | 50.55 (9.895)
  Role Emotional | 46.63 (16.00)
  Vitality | 50.47 (10.514)
  Mental Health | 51.92 (12.581)
  Physical Component Score | 46.96 (7.822)
  Mental Component Score | 50.58 (12.289)

ADVERSE EVENTS:
Time Frame: 12-months
Description: All adverse events (AEs) were coded using the Medical Dictionary of Regulatory Activities (MedDRA) Version 12.1. AEs with a definite, possible, or unable to determine relationship are considered to be related to Permacol™ surgical implant.
Arm/Group | Permacol
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Permacol (N=8)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Considered not related to procedure or device. It was later determined that the event was related to antibiotic medication.
Tachycardia (Cardiac disorders) | 1 (1) — Categorized as possibly related to Permacol™ surgical implant and procedure. The event resolved two days after onset and did not occur again throughout the study.
Cardiopulmonary Failure (Cardiac disorders) | 1 (1) — Categorized as unknown relation to procedure and no relation to device.
Left epididymal orchitis with scrotal edema (Reproductive system and breast disorders) | 1 (1) — Categorized as not related to procedure or device and was ongoing at the time of study closure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Permacol (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oropharyngeal blistering (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Adverse drug reaction (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Abdominal abscess (Infections and infestations) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Incontinence (Nervous system disorders) | 1 (1)
Urinary incontinence (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ichthyosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No